CLINICAL TRIAL: NCT04818307
Title: Long Term Effects of Mulligan Mobilization With Movement Versus Macquarie Injury Management Group on Function and Pain of Knee Osteoarthritis
Brief Title: Mulligan Mobilization With Movement Versus Macquarie Injury Management Group in Function and Pain of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/1064
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Pain; Movement with Mobilization
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Movement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Macquarie Injury Management group (Experimental)
  Interventions: Other: Macquarie Injury Management group
- Mulligan Mobilization with Movement (Active Comparator)
  Interventions: Other: Mulligan Mobilization with Movement

INTERVENTIONS:
Other: Macquarie Injury Management group — Group A was treated by MIMG (soft tissue mobilization) with base line treatment (Hot pack for 10 mint, Quadriceps Isometrics, Stretching). For the application of technique subject lies supine with extended knee, therapist places both hands on the knee and gently apply soft tissue release. This procedure was applied for 2 to 3 minutes.
  Arms: Macquarie Injury Management group
Other: Mulligan Mobilization with Movement — Group B was treated by Mulligan Mobilization with movement with base line treatment (Hot Pack for 10 mints, Quadriceps Isometrics, Stretching). For the application of technique subject lies supine with 30 degree knee flexion, therapist places right hand below the knee and left hand above the knee. Apply the lateral glide on the joint. This procedure was applied for 3 times.
  Arms: Mulligan Mobilization with Movement

SUMMARY:
Knee pain is one of the most usual pain that commonly affects people especially in the late age. It can be caused by osteoarthritis, poor posture or sitting position, bad bending or improper lifting. It is usually not caused by a serious illness. It is the most common cause of disability. To compare the long term effects of Mulligan Mobilization with Movement versus Macquarie Injury Management Group on pain and function of knee osteoarthritis.

DETAILED DESCRIPTION:
It was a randomized clinical trial conducted in Revival Physiotherapy Center, Lahore. A convenient sample of 26 diagnosed patients with osteoarthritis was included in the study. Subjects were randomly distributed in to two groups with use of flip coin method Group of randomization. Group 1 patients got MIMG with routine physical therapy and Group 2 got MWM with routine physical therapy. Visual analogue Scale (VAS),Non modified WOMAC were used to assess all patients before and after 4 weeks of intervention. Statistical analysis was computed by SPSS 20.0.

ELIGIBILITY:
Inclusion Criteria:

* ACR criteria for knee will be over age 50
* less than 30 minutes of morning stiffness,
* Crepitus on active motion,
* Tenderness
* Enlargement
* No palpable warmth of synovium.
* Osteoarthritis grade 1 and 2 by Kelly-green and Lawrence method.

Exclusion Criteria:

* Any surgical procedure done in past 6 months and metal implants in lower extremity.
* Any infection and neoplastic disorder.
* Post traumatic knee stiffness.
* Secondary knee O A peripheral vascular disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue scale | 6 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
WOMAC | 6 months
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shabbir, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kandada S, Heggannavar A. Effect of Mulligan's MWM versus Macquarie Injury Management Group (MIMG) protocol on pain and function in osteoarthritis of knee: a randomised clinical trial. IJTRR. 2015;4(4):125-31.
- [Background] Bhatia D, Bejarano T, Novo M. Current interventions in the management of knee osteoarthritis. J Pharm Bioallied Sci. 2013 Jan;5(1):30-8. doi: 10.4103/0975-7406.106561. PMID 23559821
- [Background] Felson DT. The epidemiology of knee osteoarthritis: results from the Framingham Osteoarthritis Study. Semin Arthritis Rheum. 1990 Dec;20(3 Suppl 1):42-50. doi: 10.1016/0049-0172(90)90046-i. PMID 2287948
- [Background] Felson DT, Gale DR, Elon Gale M, Niu J, Hunter DJ, Goggins J, Lavalley MP. Osteophytes and progression of knee osteoarthritis. Rheumatology (Oxford). 2005 Jan;44(1):100-4. doi: 10.1093/rheumatology/keh411. Epub 2004 Sep 20. PMID 15381791
- [Background] Cooper C, McAlindon T, Coggon D, Egger P, Dieppe P. Occupational activity and osteoarthritis of the knee. Ann Rheum Dis. 1994 Feb;53(2):90-3. doi: 10.1136/ard.53.2.90. PMID 8129467
- [Background] Alshami AM. Knee osteoarthritis related pain: a narrative review of diagnosis and treatment. Int J Health Sci (Qassim). 2014 Jan;8(1):85-104. doi: 10.12816/0006075. PMID 24899883